CLINICAL TRIAL: NCT04029467
Title: Addition of Dexmedetomidine to Ropivacaine for Ultrasound Guided Erector Spinae Block: Evaluation of Effect on Postoperative Pain After Breast Surgery: A Double-Blinded, Prospective, Randomized Clinical Trial
Brief Title: Effect of Dexmedetomidine on the Duration of Pain Control in ESP Block for Breast Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Yara Al Jalbout, Clinical Instructor, Director Anaesthesiology Residency Program, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAUMCRH.YJ1.16/Jul/2019
Record Dates: First submitted 2019-07-17; First posted 2019-07-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer; Mastectomy; Axillary Lymph Node Dissection; Pain, Postoperative
Keywords: ESP block; erector spinae plane block; mastectomy; ropivacaine; dexmedetomidine; pain; breast
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Precedex (Active Comparator): participants will receive an ESP block with 20 ml Ropivacaine 0.375% in the induction room 20 minutes before their operation
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine (Experimental): participants will receive an ESP block with 20 ml Ropivacaine 0.375% + 0.5mcg/kg dexmedetomidine in the induction room 20 minutes before their operation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — addition of dexmedetomidine to ropivacaine as an adjuvant in ESP block to assess wether or not it prolongs its duration of action

SUMMARY:
Patients undergoing Partial or total mastectomy with axillary LN dissection will receive prior to induction of general anaesthesia ESP block at T4 level at the same side of the surgery. one group will receive ropivacaine 0.375% and the other will get ropivacaine 0.375% with dexmedetomidine 0.5mcg/kg as an adjuvant. time to first narcotic requirement will be documented and therefore an assessment of the duration of action of the block will be made

DETAILED DESCRIPTION:
Background and Objective: Whether partial or complete, mastectomy with axillary lymph node dissection is a painful surgery. Acute postoperative pain management is challenging and crucial due to high chances of it transforming into chronic pain. Erector spinae plane (ESP) block has been shown to be effective in managing post mastectomy pain.Dai et al showed the effectiveness of dexmedetomidine in prolonging the duration of sensory block, motor block and analgesia when dexmedetomidine as an adjunct is added to ropivacaine in brachial plexus block (1). The aim of our study is to show the effectiveness of dexmedetomidine in prolonging the analgesic effect of ropivacaine when added to it in ESP block compared to using ropivacaine alone in patients undergoing mastectomy with axillary lymph node dissection, and to study its impact on postoperative opioid consumption.

Methods: 44 American Society of Anesthesiologist (ASA) physical status classification class I, II and III will be randomly allocated to one of two groups, both receiving a single injection erector spinae plane block at T4 vertebral level using 20ml ropivacaine 0.375% 20 minutes before the induction of anesthesia. The first group will receive 0.5mcg/kg of dexmedetomdine added to the ropivacaine solution. The control group will receive no dexmedetomidine.

Postoperatively, patients in both groups will be receive acetaminophen 1g orally every 6 hours and oxycodone 5 mg orally as needed every 6 hours if VAS is more than 4. Postoperative pain will be measured using Verbal Analogue Scale (VAS) at 0, 1, 2, 4, 6, 12, 18, and 24 hours.

Conclusion: This study will be the first of its kind to investigate the impact of adding dexmedetomidine as an adjunct to ropivacaine in prolonging the ESP block duration in patients undergoing mastectomy with axillary lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I, II and III patients
2. Age range: 18-80 years old
3. Elective partial or unilateral radical mastectomy with sentinel lymph node dissection

Exclusion Criteria:

1. Pregnant woman
2. Bilateral mastectomy.
3. Skin infection at the site of needle puncture
4. Coagulopathy problems
5. Allergy or contraindication to any of the study drugs
6. Recent use of opioid drugs

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically female
Enrollment: 44 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-07-17 (Estimated); Study Completion 2022-01-17 (Estimated)

PRIMARY OUTCOMES:
Pain assessment in the first 24 hours post operatively: VAS score | 24 hours
  Pain will be assessed using the VAS score ranging from 0, indicating no pain at all, to 10, indicating the worst pain the patient has ever felt

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese American University Medical Center-Rizk Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No